CLINICAL TRIAL: NCT04557462
Title: A Multicenter Rollover Extension Program (REP) to Evaluate the Long-term Safety and Tolerability of Open Label Iptacopan in Adult Participants With Primary IgA Nephropathy Who Have Completed Study CLNP023X2203 or CLNP023A2301
Brief Title: A Rollover Extension Program (REP) to Evaluate the Long-term Safety and Tolerability of Open Label Iptacopan/LNP023 in Participants With Primary IgA Nephropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023A2002B; 2020-002200-40 (EudraCT Number)
Expanded Access: NCT05222412 (Available)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Primary IgA Nephropathy
Keywords: Immunoglobulin A nephropathy; Primary IgA nephropathy; IgAN; chronic kidney disease; glomerulonephritis; complement alternative pathway; eGFR; UPCR; UACR; LNP023
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic; Glomerulonephritis | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LNP023 (Experimental): All participants are receiving 200 mg b.i.d
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — Capsule 200 mg (b.i.d.) taken orally twice a day
  Other Names: iptacopan

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability, of open label iptacopan in primary IgA nephropathy participants who have completed either the CLNP023X2203 or CLNP023A2301 clinical trials. The open-label design of the current study is appropriate to provide study participants the opportunity to receive treatment with iptacopan until marketing authorizations are received and the drug product becomes commercially available while enabling collection of long-term safety and tolerability data for the investigational drug. Furthermore efficacy assessments conducted every 6 months will afford the opportunity to evaluate the clinical effects of iptacopan on long-term disease progression.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multicenter roll-over extension program (REP) to:

* CLNP023X2203, a Phase II trial investigating the dose ranging effects of LNP023 on efficacy, pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability in primary IgAN patients, and
* CLNP023A2301, a Phase III trial, investigating the efficacy, pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability of LNP023 in patients with primary IgAN.

Subjects completing the CLNP023X2203 and CLNP023A2301 trials on study drug, who want to continue treatment and who meet the inclusion/exclusion requirements of the roll over extension program, will have the opportunity to receive iptacopan until:

* 3 years from LPFV of this study CLNP023A2002B, or
* the participant no longer derives benefit from iptacopan according to the Investigator, or
* the benefit-risk profile of the product in IgAN is no longer positive, or
* initiation of maintenance hemodialysis, kidney transplantation or eGFR < 15 mL/min/1.73m2 , or
* the product becomes commercially available in a specific country following product launch and subsequent reimbursement for IgAN, where applicable, or
* if a marketing application or reimbursement of an investigational product is rejected/not pursued in a region/country for the indication under study or which ever is sooner

ELIGIBILITY:
Inclusion Criteria:

* For LNP023X2203, participants must have completed part 1 or part 2 of the trial. For LNP023A2301, participants must have completed the entire core trial defined as the full 24 month treatment period.
* eGFR* ≥ 20 ml/min/1.73m2

  *eGFR calculated using the CKD-EPI formula (or modified MDRD formula according to specific ethnic groups and local practice guidelines)
* Per investigator's clinical judgement, the participant may benefit from receiving the open-label treatment of iptacopan 200 mg b.i.d.
* Prior Vaccination against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections should be up to date (i.e. any boosters required administered according to local regulations.
* All participants must be on supportive care regimen of ACEi or ARB* as per KDIGO guidelines.

  * participants who are not taking KDIGO guideline doses because they have documented allergies or intolerance to ACEi and ARB are eligible for the study

Exclusion Criteria:

* participants who screen or baseline failed in the CLNP023X2203 Part 1 or Part 2, or CLNP023A2301 studies or who prematurely withdrew from either study for any reason.
* Evidence of severe urinary obstruction or difficulty in voiding; any urinary tract disorder other than IgAN at screening and before dosing with LNP023.
* Current (within 4 weeks of study drug administration in the REP) acute kidney injury (AKI)
* Presence of Rapidly Progressive Glomerulonephritis (RPGN) as defined by 50% decline in eGFR within the last 3 months.
* Participants treated with immunosuppressive or other immunmodulatory agents such as but not limited to cyclophosphamide, rituximab, infliximab, eculizumab, canakinumab, mycophenolate mofetil (MMF) or mycophenolate sodium (MPS), cyclosporine, tacrolimus, sirolimus, everolimus and/or systemic corticosteroids exposure (>7.5 mg/d prednisone/prednisolone equivalent) within 5 half-lives of respective medication or 90 days prior to first study drug administration, whichever is shorter. Rituximab requires 180 days wash out.
* Use of other investigational drugs at the time of enrolment, or within 5 half-lives of enrolment or within 30 days whichever is longer.
* History of recurrent invasive infections caused by encapsulated organisms, such as meningococcus and pneumococcus.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2032-10-25 (Estimated); Study Completion 2032-10-25 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with serious adverse event | Date of first administration of (Day 1) to 7 days after the date of the last actual administration of study treatment
  Summary statistics on serious adverse events
Number and percentage of participants with adverse event | Date of first administration of study treatment (Day 1) to 7 days after the date of the last actual administration of study treatment
  Summary statistics on adverse events
Number and percentage of participants with adverse events of special interest | Date of first administration of study treatment (Day 1) to 7 days after the date of the last actual adminstration of study treatment
  Summary statistics on adverse events of special interest
Number and percentage of participants with abnormalities in vital signs | Date of first administration of study treatment (Day 1) to 7 days after the date of the last actual administration of study treatment
  Summary statistics on abnormalities in vital sign parameters
Number and percentage of participants with abnormalities in ECG | Date of first administration of study treatment (Day 1) to 7 days after the date of the last actual administration of study treatment
  Summary statistics in abnormalities in ECG parameters
Number and percentage of participants with abnormalities in clinical laboratory evaluations | Date of first administration of study treatment (Day 1) to 7 days after the date of the last actual administration of study treatment
  Summary statistics on abnormalities in clinical laboratory evaluations

SECONDARY OUTCOMES:
Annualized total eGFR slope | Screening visit, Months 1, 3, 6, 9, 12 and every 6 months thereafter
  Annualized rate of renal disease progression as measured by mean eGFR slope at post baseline visits
Change from baseline in eGFR | Screening visit, Months 1, 3, 6, 9, 12 and every 6 months thereafter
  Average change from baseline in eGFR at post-baseline visits
Log transformed ratio to baseline in UPCR, UACR | Screening visit, Months 1, 3, 6, 9, 12 and every 6 months thereafter
  Log transformed ratio to baseline in UPCR, UACR at post-baseline visits. The log transformation refers to the natural log (base on e)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (143):
- United States (16):
  - AZ Kidney Dise and Hypertension Ctr, Glendale, Arizona
  - Kaiser Permanente, San Diego, California
  - North America Research Institute, San Dimas, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Nephrology Associates PA, Newark, Delaware
  - CaRe Research, Chubbuck, Idaho
  - Nep Assoc of Northern Illinois, Hinsdale, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Clin Rsrch Consult a JCCT Company, Kansas City, Missouri
  - DaVita Clinical Research, Las Vegas, Nevada
  - New Jersey Kidney Care, Jersey City, New Jersey
  - Col Uni Med Center New York Presby, New York, New York
  - Dallas Renal Group, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
- Argentina (3):
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Santa Fe
- Australia (3):
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (3):
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Brazil (5):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto
- Novartis Investigative Site, Oshawa, Ontario, Canada
- Novartis Investigative Site, Temuco, Chile
- China (18):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Luoyang, Henan
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Ningbo
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenzhen
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
- Novartis Investigative Site, Prague, Czechia
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (12):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Hungary (2):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
- India (3):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
- Israel (3):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Napoli
- Japan (16):
  - Novartis Investigative Site, Kasugai, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (2):
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Querétaro
- Novartis Investigative Site, Groningen, Provincie Groningen, Netherlands
- Norway (2):
  - Novartis Investigative Site, Nordbyhagen, Oslo County
  - Novartis Investigative Site, Bergen
- Russia (2):
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Košice, Slovakia
- Slovenia (2):
  - Novartis Investigative Site, Maribor, Slovenia
  - Novartis Investigative Site, Ljubljana
- Novartis Investigative Site, Bloemfontein, Free State, South Africa
- South Korea (6):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (3):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Salamanca
- Novartis Investigative Site, Stockholm, Sweden
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Köseköy, Kocaeli
  - Novartis Investigative Site, Antalya, Konyaalti
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Istanbul, Sariyer
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
- United Kingdom (5):
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Salford
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.